CLINICAL TRIAL: NCT05959746
Title: Clinical Development of a Tool for Optimized Self- and Hetero-diagnosis of Stroke Using Artificial Intelligence: Stage1- Collection of Video-clinical Data in a Pragmatic Situation.
Acronym: PREDISTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Société par Action Simplifiée AI-Stroke (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIVI/2022/ET-01
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Stroke, Cerebrovascular
Keywords: Artificial Intelligence; Data bank; Video recording
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with suspected acute stroke (Experimental)
  Interventions: Other: AI-STROKE application

INTERVENTIONS:
Other: AI-STROKE application — Complete neurological exam of stroke patients will be filmed by healthcare workers and themselves using the AI-STROKE application

SUMMARY:
The study authors aim to form a collection of video-clinical data in a pragmatic situation to enable the development of relevant AI algorithms (for both hetero- and self-diagnosis modes). The aim is to optimize management through early diagnosis (self- and hetero-diagnosis) and thus to reduce sequelae disability.

The study authors hypothesize that some stroke patients will be able to successfully perform a self-test consisting of a few exercises dictated by an application on a smartphone or tablet and recorded on video.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in the emergency department or hospitalized in the NICU at the CHU de Nîmes for suspected stroke or transient ischemic attack in the acute phase (<72h), with or without motor deficit
* Patient to be seen again in consultation within 4 months
* Patient has given free and informed consent and signed the consent form. If the patient is not in a position to give consent, it must be obtained, prior to filming the first video, from the designated trusted support person or relatives present. In this case, data will not be used until the patient is able to sign the consent (CNIL).
* Patient affiliated or beneficiary of a health insurance scheme

Exclusion Criteria:

* Patients who do not speak or read French.
* Patient in a period of exclusion determined by another study.
* Patient under court protection, guardianship or curatorship.
* Pregnant, parturient or breast-feeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Usable video recording made by the patient | Day 0
  Recording using AI-STROKE application
Usable video recording made by the hospital worker | Day 0
  Recording using AI-STROKE application

SECONDARY OUTCOMES:
Usable video recording made by the patient | Month 3
  Recording using AI-STROKE application
Usable video recording made by the hospital worker | Month 3
  Recording using AI-STROKE application
Feasibility of patient self-recording | Day 0
  Patient able to record without assistance: yes/no
Feasibility of patient self-recording | Month 3
  Patient able to record without assistance: yes/no
Acceptability of self-recording by patients | Month 3
  Patient accepting to self-record: Yes/no
Patient-reported ease of self-recording | Day 0
  Visual numerical scale 0-10
Patient-reported ease of self-recording | Month 3
  Visual numerical scale 0-10
Stroke severity | Day 0
  NIHSS (National Institute of Health Stroke Scale) score assessed by neurologist
Stroke severity | Month 3
  NIHSS (National Institute of Health Stroke Scale) score assessed by neurologist
Degree of disability following stroke | Day 0
  mRS (modified Rankin Scale) score, range 0 (no symptoms) to 5 (severe handicap) administered by the neurologist
Degree of disability following stroke | Month 3
  mRS (modified Rankin Scale) score, range 0 (no symptoms) to 5 (severe handicap) administered by the neurologist

CONTACTS AND LOCATIONS:
Overall Officials: Anne WACONGNE, Principal Investigator — CHU de Nimes
Locations (1):
- Centre Hospitalier Universitaire, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No